CLINICAL TRIAL: NCT01572688
Title: A Multicenter, Single Arm, Open Label Study of Autologous Stem Cell Transplantation With High Dose Melphalan in Patients With Multiple Myeloma
Brief Title: Safety and Efficacy Study of High Dose Melphalan to Treat Multiple Myeloma
Acronym: MM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Lanjin Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG0276
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous stem cell transplant (Experimental)
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — powder for injection, 200mg/m2, uses after reconstituted within 24 hours

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of melphalan for injection for autologous stem cell transplant in multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Patients with greater or equal to 18 years, with a upper age limit of 65 years are eligible.
* Multiple myeloma patients, symptoms conform to diagnosis of multiple myeloma of IMWG2003/WHO2008 criteria.
* Patients with responsive disease after induction therapy not more than 6 courses of treatment
* A complete response
* A very good partial response
* A partial response
* At least 4 weeks long from last cytotoxic treatment(exclude Bortezomib, thalidomide, dexamethasone);
* Eastern Cooperative Oncology Group (ECOG) scored 0 or 1 Patient has an absolute neutrophil count of ≥1.5×109/L and platelet count≥80×109/L;
* Calculated creatinine clearance >50ml/min by Cockcroft-Gault formula or collect urine within 24 hours.
* Patient with a total bilirubin ≤1.5 times of normal upper limit, AST,ALT≤2.5times of normal upper limit;
* Cardio-pulmonary function is adequate to conduct autologous stem cell transplant.
* Ratio of body weight and ideal body weight <175%;
* All patients should have a life expectancy of more than 12 weeks
* Signed informed consent form voluntarily

Exclusion Criteria:

* CD34 positive hematopoietic stem cell collected <2.0×106/kg
* Patients have a psychiatric history
* Female subject is pregnant or breast-feeding
* Patients are hypersensitive to this trial product or other alkylating agents
* Participate of other clinical trials within the past 4 weeks Active CNS lesions
* Concomitant of active infection or positive of HIV antibody
* Concomitant of other un-healed malignancy
* Left ventricular ejection fraction≤50%
* Patients with serious thrombosis
* Any severe concomitant disease that will expose study subjects to unacceptable risks.
* Patients not suitable to enroll by investigators considerations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
1 year Progression Free Survival | 20 months
  Plan to enroll all trial subjects within 8 months and follow up 1 year for each subject after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, master, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Hematologic Hospital of Chinese Academy of Medical Sciences, Tianjin, China